CLINICAL TRIAL: NCT01356537
Title: Non Interventional Study of VPRIV® (Velaglucerase Alfa) Home Therapy in Patients With Gaucher's Disease
Brief Title: Home Therapy With VPRIV in Gaucher's Disease
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: Shire/CS03
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gaucher's Disease under VPRIV

SUMMARY:
The purpose of this study is to proof increasing patient satisfaction and preservation of quality of life in patients with Gaucher's Disease receiving their enzyme replacement therapy with VPRIV (Velaglucerase alfa)at their home setting compared to receiving the infusions at the clinic or at doctor's practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a confirmed diagnosis of Gaucher disease type 1
* Age> 2 years
* patients who have at least 3 infusions (6 weeks) at least 5-year or 5-6 infusions (10-12 weeks) at 2 - to 4-year patients have received VPRIV ® and tolerate well
* The patient is compliant, the previous VPRIV ® infusions were / performed approximately every 2 weeks in the center during office visits
* The patient was already before inclusion in this study for a home infusion therapy and has consented to (or their legal representative)
* The patient / be lawful. Representative has consented in writing to participate in this study.

Exclusion criteria:

• The patient is participating in a clinical trial with a medicinal product

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proven Gaucher's Disease foreseen for home treatment with VPRIV (Velaglucerase alfa) at German Gaucher centers
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-05-20 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction estimated on a 10-ary Likert scale, quality of life estimated by SF-36 questionnaire | comparison of baseline to 12 months value

SECONDARY OUTCOMES:
Number (per infusion) and severity of infusion-related side effects | baseline compared to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Austria (5):
  - Landeskrankenhaus Bregenz, Bregenz
  - Paracelsus Medizinische Privatuniversität Salzburg, Salzburg
  - AKH, Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Medical University of Vienna, Vienna
  - Medizinische Universität Wien, Vienna
- Germany (6):
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Cologne
  - Universitätsklinikum Mainz, Mainz
  - Klinikum rechts der Isar, München
  - Albrecht-Kossel-Institut für Neuroregeneration (AKos), Rostock
  - Helios Klinikum Schwerin, Schwerin
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fd24db2bf003ab46aa1